CLINICAL TRIAL: NCT02409030
Title: Validation Trial for a Multi-parameter Diagnostic Blood Test for the Diagnosis of Alzheimer's Disease
Brief Title: Multi-parameter Diagnostic Blood Test for the Diagnosis of Alzheimer's Disease
Acronym: RH-VAL
Status: Completed | Type: Observational
Sponsor: Raman Health Technologies, S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: RH-VAL-2013-01
Record Dates: First submitted 2015-03-17; First posted 2015-04-06 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 tubes of blood ( 30 mL of blood in total) for further analysis of their products (plasma, cells and DNA) in Alzheimer's research unit project CIEN Foundation would be extracted .
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cognitively Healthy controls: The neuropsychological test assessment must confirm that there is no cognitive impairment.
  In the case of the cognitively healthy controls, CerebroSpinal Fluid tests performed within 24 months of inclusion will be accepted.
- Alzheimer Disease: Patients with AD will be classified based on currently valid and updated diagnostic algorithms in the NIA-Alzheimer's Association of America Clinical Guidelines (2011).
- Frontotemporal dementia: Inclusion criterion used will be prior diagnosis based on the diagnostic guidelines published by Dr. Rackovsky (Brain, 2011) for the behavioural variant; and those published by Prof. D. Neary (Neurology, 1998) for primary aphasia. A clinical and neuropsychological assessment is required, with the optional presence of alterations to the progranulin gene (and others) and there must be a compatible, previously performed imaging test (MRI, PET or SPECT) (predominantly frontal or frontotemporal atrophy).

SUMMARY:
The purpose of this study is to validate a diagnostic test that combines different blood markers to identify and correctly classify patients with Alzheimer's disease (AD) compared to individuals with behavioural variant frontotemporal dementia (bvFTD, patient control) versus cognitively healthy individuals (healthy control).

DETAILED DESCRIPTION:
The purpose of this study is to validate a new multi-parameter diagnostic test, on a well-characterised population based on new AD diagnostic criteria, that combines different types of markers, selected based on prior exploratory studies carried out by Raman Health Technologies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls:

   * Aged between 50-80 years.
   * Men and women.
   * Assessment of the neuropsychological tests confirming the absence of cognitive impairment.
   * Prior to participant inclusion, obtaining the results of the CerebroSpinal Fluid marker analysis (beta-amyloid, Tau protein and p-Tau) carried out in the 24 months before recruitment.
2. Patients diagnosed with Alzheimer's disease (AD).

   * Aged between 50-80 years.
   * Men and women.
   * Patients meet the clinical criteria for Alzheimer's disease:
   * Prior to participant inclusion, results obtained from CerebroSpinal Fluid marker analysis (beta-amyloid, Tau protein and p-Tau) carried out in the 36 months before recruitment.
3. Patients with behavioural variant frontotemporal dementia and primary progressive aphasia: -

   * Aged between 50-80 years.
   * Men and women.
   * Patient meets the clinical criteria of behavioural variant frontotemporal dementia (bvFTD), or syndromes associated with temporal variants that affect language (primary progressive aphasia, agrammatic and semantic subgroups):

(Mild Cognitive Impairment) sub-study: Patients with mild cognitive impairment will be included

* Aged between 50-80 years.
* Men and women.
* Patient meets the clinical criteria for mild cognitive impairment:
* Clinical diagnostic criteria for mild cognitive impairment: NIA-Alzheimer's Association of America criteria, Alzheimer's Dementia, 2011
* Prior to participant inclusion, results obtained from cerebrospinal fluid marker analysis (beta-amyloid, Tau protein and p-Tau) carried out in the 12 months before recruitment.

Exclusion Criteria:

* Severe or acute systemic disease that could impede the participant's follow-up study: Advanced liver or kidney disease and disseminated neoplastic disease
* Addiction to alcohol or other drugs in the last two years based on Diagnostic and Statistical Manual of Mental Disorders IV criteria, except nicotine use, which is permitted
* Down's syndrome
* Moderate or severe head injury
* central nervous system infections (HIV, syphilis, borrelia, herpes simplex, suspected Creutzfeldt-Jakob disease)
* Endocrine alterations (thyroid alterations)
* Nutritional deficiency (vitamin B12, folic acid)
* Clinical history of stroke in the previous three months or neuroimaging evidence of clinically significant cardiovascular disease (e.g. strategic infarct or severe leukoencephalopathy).
* Neurological diseases (dysmyelinating disorders, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, subdural haematoma, brain tumours)
* Major psychiatric disorder (major depression or psychosis)
* Patients who do not have a clearly defined clinical diagnosis according to the study groups (inclusion/exclusion criteria)
* Disease which, in the investigator's or sponsor's judgement, may have a potentially significant influence and thus generate bias in the study markers.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is estimated that a sample of 500 patients (250 with AD and 250 with FTD) and 200 controls (700 individuals in total) will be sufficient to corroborate the hypothesis that permits validation of the new diagnostic test. The sample size estimate is based on a hypothesis of non inferiority between the new test and the test used in normal clinical practice, expecting a 10% delta of the 75% validity, sensitivity and specificity indices with an alpha error of 0.05 and a beta error of 0.20.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Blood markers | Up to 12 months
  Multi-parameter determination: Raman laser and infrared spectroscopic markers, Metabolite-based markers (A02, A16, A22 ST01 F20 M30), Protein markers (A, A-T, B, PRO-B, C, C1, C2, PROGRANULIN), Biochemical markers (OXIDATIVE STRESS MARKERS, CTAN, ROUTINE BIOCHEMICAL MARKERS (GLUCOSE, TRIGLYCERIDES) and Genetic markers (ApoE, ApoC).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cabello, Study Director — Raman Health Technologies, S.L.
Locations (16):
- Belgium (2):
  - AZ Sint Jan, Bruges
  - UCL St Luc, Brussels
- France (5):
  - Centre Hospitalier d'ARRAS, Arras
  - Hôpital neurologique Pierre Wertheimer, Bron
  - Clinique Neurologique CHRU, Lille
  - Centre Mémoire paris Nord Ile de France GH Saint-Louis Lariboisière Fernand Widal, Paris
  - Cognitive and Behavioral Disease Center and Alzheimer's Institute, Paris
- Spain (9):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - CITA Alzheimer, Donostia / San Sebastian, San Sebastián
  - Hospital Sant Pau, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided